CLINICAL TRIAL: NCT04243070
Title: Collection of ECG Signals From Various Patient Groups for the Development of Algorithms for Sensing and Detection of Rhythm Anomalies
Brief Title: BIO|CONCEPT.ECG-Library (Collection of ECG Signals for Development of Algorithms)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment rates so that proper completion of the study cannot be expected anymore.
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RD023
Record Dates: First submitted 2020-01-24; First posted 2020-01-27 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-08

CONDITIONS: Heart Diseases; Rhythm; Abnormal
Keywords: Holter ECG recording
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-channel Holter ECG recording for EPS patient (Other): Patients participating in an EPS will undergo a 3-channel Holter ECG recording in parallel to the standard 12-channel Holter ECG recording during the EPS followed by an optional 24 h observation period
  Interventions: Diagnostic Test: 3-channel Holter ECG recording
- 12-channel Holter ECG recording for non-EPS patients (Other): Patients scheduled for a follow-up for their heart disease will undergo a 12-channel Holter ECG recording while participating in a Body Motion test followed by a 24 h observation period
  Interventions: Diagnostic Test: 12-channel Holter ECG recording

INTERVENTIONS:
Diagnostic Test: 3-channel Holter ECG recording — 3-channel Holter ECG recording for patients undergoing an EPS
  Arms: 3-channel Holter ECG recording for EPS patient
Diagnostic Test: 12-channel Holter ECG recording — 12-channel Holter ECG recording for patients undergoing a routine follow-up
  Arms: 12-channel Holter ECG recording for non-EPS patients

SUMMARY:
Collection of Holter surface ECGs for the development of new sensing and detection algorithms

DETAILED DESCRIPTION:
The aim of the study is to collect data from surface ECGs by using Holter ECG recordings from patients with different forms of diagnosed arrhythmias and/or specific ECG characteristics from heart diseases to support the development of new sensing and detection algorithms for implants.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to understand the nature of the study and willing to provide written informed consent.
* Patient is willing and able to attend Holter ECG procedure following a visit
* History of at least one of the following conditions (established via ECG prior to enrollment):

(A) Patient with pacemaker/ICD and

1. Ventricular stimulation > 30 % or

   (B) Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and at least one of the following:
2. Frequent Ventricular Extrasystoles (VES) (incl. Bigeminus) or
3. Atrioventricular Reentrant Tachycardia (AVRT)/Wolff-Parkinson-White (WPW) syndrome or
4. Atrioventricular Nodal Reentrant Tachycardia (AVNRT) or
5. Sinus Tachycardia at rest or
6. Atrial Flutter or
7. Any form of Ventricular Tachycardia (VT) or
8. Silent/Paroxysmal/persistent/permanent AF or
9. Brugada syndrome or
10. Long QT syndrome or
11. Right Bundle Branch Block (RBBB) or
12. Left Bundle Branch Block (LBBB) or
13. Myocardial Ischemia/Acute Myocardial Infarction or
14. Other abnormal QRS(T) complex, ST segment or T-wave morphology, i.e. any other QRS anomaly / ST segment elevation / ST segment Depression / T wave changes

Exclusion Criteria:

* Any condition which precludes the patient's ability to comply with the study requirements.
* Known allergy to patch electrodes.
* Pregnant or breast feeding.
* Less than 18 years old.
* Participation in another interventional clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Contzen, Dr., Study Chair — Biotronik SE & Co. KG
Locations (5):
- Germany (5):
  - Vivantes-Krankenhaus im Friedrichshain, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Gießen und Marburg GmbH (UKGM), Giessen
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3-channel Holter ECG Recording for EPS Patient | 12-channel Holter ECG Recording for Non-EPS Patients
Started | 66 | 23
Completed | 66 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: According to the statistical analysis plan it was pre-specified to report baseline data for the total population only.
Arm/Group | Total
Number analyzed (Participants) | 89
Age, Continuous [Median (Standard Deviation); unit: years] | 64.0 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 89

OUTCOME MEASURES:

1. Primary Outcome: Number of Successful ECG Recordings Per Condition
Description: All ECG recordings were evaluated by an internal board and all patients were allocated to one of 15 groups (covering 14 ECG patterns of interest and one group for "no ECG pattern of interest recorded").
Time Frame: 24 hours
Population: According to the statistical analysis plan it was pre-specified to report the number of successful Holter recordings per ECG pattern for all patients irrespective of the method for Holter recording.
Measure: Number; unit: Successful ECG recordings
Units Other Than Participants: Holter ECG recordings
Groups:
- Patient With Pacemaker/ICD and Vp > 30%: Patient with pacemaker/ICD and Ventricular stimulation > 30 %
- Frequent Ventricular Extrasystoles (VES) (Incl. Bigeminus): Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and 2. Frequent Ventricular Extrasystoles (VES) (incl. Bigeminus)
- Atrioventricular Reentrant Tachycardia (AVRT)/Wolff-Parkinson-White (WPW) Syndrome: Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and Atrioventricular Reentrant Tachycardia (AVRT)/Wolff-Parkinson-White (WPW) syndrome
- Atrioventricular Nodal Reentrant Tachycardia (AVNRT): Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and Atrioventricular Nodal Reentrant Tachycardia (AVNRT)
- Sinus Tachycardia at Rest: Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and Sinus Tachycardia at rest
- Atrial Flutter: Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and Atrial Flutter
- Any Form of Ventricular Tachycardia: Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and any form of Ventricular Tachycardia
- Silent/ Paroxysmal/ Persistent/ Permanent Atrial Fibrillation (AF): Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and silent/ paroxysmal/ persistent/ permanent Atrial Fibrillation (AF)
- Brugada Syndrome: Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and Brugada syndrome
- Long QT Syndrome: Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and Long QT syndrome
- Right Bundle Branch Block (RBB): Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and Right Bundle Branch Block (RBB)
- Left Bundle Branch Block (LBB): Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and Left Bundle Branch Block (LBB)
- Myocardial Ischemia/ Acute Myocardial Infarction: Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and Myocardial Ischemia/ Acute Myocardial Infarction
- Other Abnormal QRS(T) Complex, ST Segment or T-wave Morphology: Patient either without pacemaker/ICD or with pacemaker/ICD, but without significant atrial and ventricular stimulation and other abnormal QRS(T) complex, ST segment or T-wave morphology
- No ECG Pattern of Interest Recorded: Patient with no ECG pattern of interest recorded
Arm/Group | Patient With Pacemaker/ICD and Vp > 30% | Frequent Ventricular Extrasystoles (VES) (Incl. Bigeminus) | Atrioventricular Reentrant Tachycardia (AVRT)/Wolff-Parkinson-White (WPW) Syndrome | Atrioventricular Nodal Reentrant Tachycardia (AVNRT) | Sinus Tachycardia at Rest | Atrial Flutter | Any Form of Ventricular Tachycardia | Silent/ Paroxysmal/ Persistent/ Permanent Atrial Fibrillation (AF) | Brugada Syndrome | Long QT Syndrome | Right Bundle Branch Block (RBB) | Left Bundle Branch Block (LBB) | Myocardial Ischemia/ Acute Myocardial Infarction | Other Abnormal QRS(T) Complex, ST Segment or T-wave Morphology | No ECG Pattern of Interest Recorded
Number analyzed (Participants) | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89
Number analyzed (Holter ECG recordings) | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89 | 89
Successful ECG recordings | 6 | 12 | 4 | 7 | 7 | 8 | 11 | 10 | 3 | 0 | 5 | 5 | 3 | 4 | 4

ADVERSE EVENTS:
Time Frame: 2 days on average
Arm/Group | 3-channel Holter ECG Recording for EPS Patient | 12-channel Holter ECG Recording for Non-EPS Patients
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/23
Serious Adverse Events (participants affected / at risk) | 3/66 | 0/23
Other Adverse Events (participants affected / at risk) | 1/66 | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3-channel Holter ECG Recording for EPS Patient (N=66) | 12-channel Holter ECG Recording for Non-EPS Patients (N=23)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | NA
Pericardial effusion (Cardiac disorders) | 2 (2) | NA
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3-channel Holter ECG Recording for EPS Patient (N=66) | 12-channel Holter ECG Recording for Non-EPS Patients (N=23)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bone marrow infiltration (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Endometrial disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Puncture site haematoma (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT04243070/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT04243070/SAP_001.pdf